CLINICAL TRIAL: NCT05101239
Title: Acute and Mild Traumatic Brain Injury in a Military (and Civilian) Population Using Advanced Microstructure Imaging in Novel Ultra-High Performance MRI
Brief Title: Acute and Mild TBI Injury in Military and Civilian Population Using Advanced MR Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: The Geneva Foundation (Other)
Collaborators: General Electric (Industry); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vincent B Ho, Director of Research, Department of Radiology, Walter Reed National Military Medical Center
Other Study IDs: 11123-0001-0001-0206
Record Dates: First submitted 2021-10-14; First posted 2021-11-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Mild Traumatic Brain Injury
Keywords: MRI; DTI; Enhanced; MR; Gradients; mTBI
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- A: Acute mTBI: Consists of up to 80 patients with acute mTBI. All acute mTBI subjects will be scanned per the HHI study design at 3 to 5 timepoints relative to their time of injury ( Visit 1 within 72 hours; Visit 2, 7 +/- 4 days; Visit 3, 30 +/- 7 days; Visit 4, 90 +/- 14 days; Visit 5, 180 +/- 30 days from injury). Even though for practicality Visits 1 and 5 are optional, every effort will be made to image as close to the time of acute injury as possible and to complete imaging for all time points.
  Interventions: Device: MRI imaging exam
- B: Control: Consists of 40 age-matched participants described above who will undergo imaging twice on the MAGNUS 3.0T MRI scanner at two distinct time points. The 2 MRI imaging sessions will be at least 2 weeks apart. One of the 2 visits will include a clinical MRI scan using the same MRI acquisition protocols used for Group A. Because age-matched Controls are not expected to exhibit structural and functional changes during the study period, it was not deemed necessary for the interval between scan-visit time points to be identical for all participants in Group B.
  Interventions: Device: MRI imaging exam
- C: Chronic mTBI: Consists of 40 age-matched participants with chronic mTBI (≥6 months and <5 years from mTBI injury to enrollment). Participants in this group will have 1 set of procedures at the Baseline Visit. This cohort will be used to understand functional and structural changes in chronic mTBI patients to identify indications of progression of patients from the acute to chronic phase
  Interventions: Device: MRI imaging exam

INTERVENTIONS:
Device: MRI imaging exam — 3T MRI scan using with ultra high performance gradient subsystem (MAGNUS MRI)

SUMMARY:
This is a prospective longitudinal study of patients with acute mTBI and comparison with chronic mTBI patients and a cohort without history of TBI or none within 5 years of enrollment. The patients will be recruited from the eligible population at military medical centers in the National Capital Region.

DETAILED DESCRIPTION:
All patients seen with suspected mTBI will undergo standard TBI assessment per institutional standard operating procedure. Mild TBI will be defined by Department of Defense/Department of Veterans Affairs Consensus- based Classification of Closed TBI Severity. This project will leverage several existing TBI clinics/programs and benefits from the clinical and technical knowledge gained from each. All participants will undergo the same screening, eligibility assessment, informed consent, baseline history/physical, statement of negative pregnancy status (if applicable), survey questionnaires, VOMS, BESS, King-Devick and abbreviated neurocognitive testing once. Participants will undergo research MRI twice at time points > 2 weeks apart and one clinical MRI. Blood samples will be collected at each study visit. The research blood specimens will be processed immediately, frozen and sent to the WRNMMC Research Laboratory for future biomarker and genomic analysis.

MRI imaging findings (common data elements or newer imaging biomarkers discovered during the initial two-year technical development phase) will be analyzed to determine the most relevant biomarkers indicative of mTBI injury and/or prognosis for recovery. More advanced correlation analysis and relative risk regression will be performed to correlate mTBI and PTSD and their comorbid associations (e.g., depression, anxiety), Statistical tests will be corrected for multiple comparisons as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Group A (acute mTBI) Adult (ages 18-55 years) any gender, who is capable of giving informed consent, having neurocognitive testing and questionnaires, able to undergo MRI, and willing to attend at least 3 of the 5 proposed clinic visits at WRNMMC.

  * Has a mild traumatic brain injury for which the individual sought medical attention in an ED/acute care clinic within 72 hours of injury.
  * Diagnosis of mTBI Acute injury and able to enroll in the study within 11 days from injury.
* Group B (Control) Adult (18 to 55 years), any gender, who is capable of undergoing informed consent, having neurocognitive testing and questionnaires, able to undergo MRI, and able to go to WRNMMC for imaging.

  * Has not had a mild traumatic brain injury in the last 5 years or ever.
* Group C (chronic mTBI) Adult (18 to 55 years), any gender, who is able to undergo MRI, and able to go to WRNMMC for imaging, capable of giving informed consent, and having neurocognitive testing and questionnaires.

  * Injury greater than 6 months but fewer than 5 years ago.

Exclusion Criteria:

* Groups A,B,C: Patients with contraindication to MRI (per standard WRNMMC SOP these individuals will not be scanned anyway. Standard WRNMMC MR screening criteria will be used as a part of their normal MR examination- e.g. non-FDA approved pacemakers, aneurysm clips,MR contraindicated metal/metallic devices, etc.).
* Groups A,B,C: Never had a penetrating, moderate or severe TBI at any time.
* Groups A,B,C: Unable to tolerate proposed imaging (e.g. severe claustrophobia, unable to tolerate lying flat for duration of MRI).
* Groups A,B,C: History of pre-existing neurologic condition which would affect the ability to interpret MRI results (such as prior stroke, multiple sclerosis, or brain tumor).
* Groups A,B,C: Patients requiring anesthesia support for sedation
* Groups A,B,C: Pregnant patients
* Groups A,B,C: Any person who is unable to sign/give consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: DoD beneficiary population
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
1. To identify objective imaging biomarkers (distinctive imaging findings) that are indicative of acute mTBI using the proposed advanced MAGNUS 3T MRI system designed for brain assessment | 6 months
  Imaging biomarkers identified on MAGNUS MRI in patients with acute mTBI
2. To identify novel and/or improved imaging biomarkers in patients with chronic mTBI (≥6 months) using the MAGNUS 3T MRI system | Up to 5 days
  Imaging biomarkers on MAGNUS MRI in patients with chronic mTBI
3. To compare images from the MAGNUS 3T MRI system to the convention 750 3T MRI system | Up to 2 weeks
  Imaging biomarkers identified on MAGNUS MRI but not on traditional MRI imaging exam

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Foo, PhD, Principal Investigator — General Electric Research
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia